CLINICAL TRIAL: NCT00376155
Title: Comparison of Two Strategies for the Delivery of Intermittent Preventive Treatment in Children (IPTc) in an Area of Seasonal Malaria Transmission
Brief Title: Comparison of Two Strategies for the Delivery of IPTc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITCRVG47; SCC990
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Malaria
Keywords: malaria; prevention; intermittent; drugs
MeSH Terms: conditions — Malaria | interventions — Sulfadoxine; Pyrimethamine; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sulfadoxine /pyrimethamine plus amodiaquine

SUMMARY:
Antimalarial chemoprophylaxis can reduce morbidity and mortality from malaria in children. However, this approach to malaria control has not been implemented widely because of concerns over its possible effect on the development of resistance and natural immunity. Intermittent preventive treatment (IPT) may be able to achieve some of the beneficial effects of chemoprophylaxis without its drawbacks. Recently, it has been shown that IPT given to Senegalese children under the age of five years on three occasions during the malaria transmission season reduced the incidence of clinical malaria by approximately 90%. However, it is uncertain how this intervention can be most effectively delivered. Therefore, 26 Maternal and Child Health (MCH) trekking clinics in Upper River Division, south of the River Gambia, each with an average catchment population of 400-500 children under 5 years of age, will be randomly allocated to receive IPT from the MCH trekking team or from a IPT dispenser (village health worker, traditional birth attendant or a community mother based in a primary health care village). Treatment with a single dose of sulfadoxine /pyrimethamine (SP) plus three doses of amodiaquine will be given to all study subjects at monthly intervals on three occasions during the months of September, October and November. The primary end points will be the incidence of clinical attacks of malaria detected by passive case detection, and cost-effectiveness of the delivery methods. Important secondary endpoints will be the coverage and the equity of coverage of IPT in preventing malaria morbidity.

DETAILED DESCRIPTION:
3. OBJECTIVES

The objective of this trial is to study the effectiveness and cost-effectiveness of two approaches to the administration of intermittent preventive treatment to Gambian children - distribution by village volunteers or through EPI trekking teams.

5 STUDY DESIGN AND METHODOLOGY

The unit of randomization will be the catchment population of the monthly EPI trekking clinics. There are 33 trekking clinics in total on the south bank of URD of which 27 are rural. The rural trekking clinics will be selected for randomization. 26 rural clusters (two will be merged to give an even number) will be stratified by health facility catchment area (Gambissara, Basse, Fatoto). Constrained randomization will be used to ensure balance within strata with regard to distribution of PHC key villages and population size.

The bednet coverage in URD is estimated to 65%. However, during the enumeration, details of bed net usage by the community will be assessed. In collaboration with the malaria control programme, we will facilitate the provision of bed nets to households without one. At the beginning of the rainy season permethrin will be provided to all households with bednets.

5.1 Malaria card

After the enumeration has been completed, a database containing the list of eligible children will be established. The database will be used to generate the list of participating study children in each village. A record system using appropriate visual aids will be devised that can be used by an IPTc dispenser. This will consist of a "malaria card" held by the mother or guardian of each child and an IPT register held by IPTc dispenser or staff of the DHT trekking team. On the malaria card held by the mother, the compound number and study number will be written in Arabic and English, together with the child's name and the name of his or her parents. The dosage of trial medication to be given will be indicated on the malaria card and the register using coloured circles and semi-circles (full circle for one tablet and semi-circle for half a tablet). The register held by the IPTc dispenser or DHT staff will contain similar information to that on the malaria card.

When a child presents to a health facility for medication, the DHT staff or the IPTc dispenser will examine the malaria card of the study subject. Medication will only be given to study subjects after correct identification and after matching the information on the malaria card held by the mother and that on the register held by the IPTc dispenser or the DHT. It is envisaged that the DHT staff and IPTc dispenser taking part in the study will be paid modest salary supplements for their contribution to the project. However, the details of payment will be discussed with the EPI unit and Basse DHT.

5.2 Cross-section survey

In December, at the end of the malaria transmission season, a cross-sectional survey of children less than 6yrs will be undertaken in all the 26 clusters. A questionnaire to determine asset rating and wealth index will be completed. Information on demographic, bed net usage, socio-economic status, health seeking behaviour and utilisation patterns profiles will be collected, a clinical history will be obtained and a physical examination will be performed, including abdominal palpation for splenomegaly and measurement of height, weight and axillary body temperature.

5.3 Distribution of tablets

5.3.1 Distribution of tablets in the villages

Each key PHC village has a health post staffed by a community health nurse. There are 29 PHC villages and the majority of these have a village health worker and a traditional birth attendant. The three towns with basic health facilities (Basse, Fatoto and Gambisara) will be excluded from the evaluation, and the trial will focus on other communities in the study area. The trial medication will be administered by IPTc dispenser based in a PHC village. The IPTc dispenser will distribute the trial medication at a central point (usually a health post) on the first Wednesday of the month during September, October and November. Mothers and carers will be asked to bring their children to the central point during the morning when the IPTc dispenser will be available to distribute the drugs. When a child presents to the central point for medication, the IPTc dispenser will identify the study subject using the malaria card held by the mother and match the information on the malaria card with that on her register. When she is satisfied that she has correctly identify the study subject and that the information on the malaria card matches those on her register, the correct dosage of the trial medication will be given to the study subject.

The first dose of treatment will be taken under direct supervision of the IPTc dispenser and she will mark her register and the malaria card to show that the child has received the tablets. The remaining two doses will be given to the mother or guardian of the child with clear instructions on how to administer the drugs.

5.3.2 Distribution of tablets in the trekking clinics A member of the MCH trekking team (designated as an IPTc officer) of each of the 3 basic health facilities (Basse, Fatoto and Gambissara) will be identified by the EPI team and given responsibility for delivery of IPT at the trekking clinics, which are allocated by randomization to deliver IPTc. Thus, each EPI team will deliver IPTc in some of its trekking clinics but not in others.

The dates of each monthly treatment will be written in Arabic and English on the "malaria cards". To ensure that children do not receive more doses of IPTc than they should, different coloured "malaria cards" will be issued to children in villages where children will receive their medication from IPTc dispenser and to those allocated to receive medication from the MCH trekking clinic. IPTc dispensers and IPTc officers will be taught how to give medication only to children who have the correct coloured cards.

At the end of the malaria transmission season, the total number of complete treatment doses each child in the trial has taken will be recorded. Compliance will be checked on a rolling basis throughout the study by assessing the number of correct doses of medication received. In addition, urine samples will be collected from a random sample of 100 children each month in the two-week period following administration of IPTc to test for the presence of SP in the urine using Eggelte dipsticks.

5.4 Morbidity surveillance during the rainy season

Passive surveillance for malaria will be maintained throughout the transmission season.

5.5 Surveillance for severe malaria

Records will be kept of admission of study children to Basse and Fatoto Health Centres. Physicians and nurses based at these facilities will be asked to look out for any child with severe malaria, and any admission attributed to malaria will be carefully documented.

5.6 Surveillance for overall and cause specific mortality

Deaths will be investigated using postmortem questionnaire techniques and cause of death established wherever possible.

5.7 Nested case control study

To estimate the effect of inequalities in wealth on malaria morbidity and its prevention by intermittent treatment, -a nested case control approach will be used to determine distribution of malaria morbidity in relation to two measures of socioeconomic status - a wealth rating scale and an asset index.

5.8 Study of cost-effectiveness

A cost-effectiveness analysis will be undertaken from a societal perspective, meaning that all costs and effects, no matter to whom they accrue, will be measured and valued.

5.8.1 Programme costs:

The costs of the two modes of delivering IPTc will be assessed using the bottom-up or 'ingredients' approach which involves the identification of all the resources required by the two modes of delivery.

5.8.2 Resource savings:

The modes of delivery will be compared with respect to the resource savings resulting from fewer children being treated for malaria related illnesses as a result of better IPTc coverage.

5.8.3 Cost-effectiveness:

For both modes of delivery, two cost-effectiveness ratios will be calculated: (i) cost per child who fully adheres to treatment; (ii) cost per case of malaria averted. In addition, net cost-effectiveness ratios will be calculated by subtracting resources saved from the total programme cost divided by the relevant outcome measure. The incidence of malaria and the costs will be compared between the two delivery arms and the cost per additional case averted calculated.

5.9 Equity

The impact of the different delivery strategies on alleviating (or exacerbating) three forms of equity will be measured. Equity outcomes and the cost of each delivery mode will also be compared using benefit-incidence analysis.

5.9.1 Equality of utilization or adherence:

To determine impact in terms of IPT coverage, levels of adherence will also be compared across the two delivery strategies; a cross-section survey will be used.

5.9.2 Equality of access:

Here we are measuring whether households have the same opportunity to benefit from each mode of delivery. This involves defining and measuring financial access, geographical access, informational access and cultural/gender barriers to access. Approximately 25 compliers and 25 non-compliers from a sub-sample of 12 clusters will be interviewed about factors influencing access to each delivery strategy.

5.9.3 Benefit-incidence-analysis:

Utilization and access data for rich and poor households will be compared with the cost of providing the service. This will involve the use of benefit-incidence-analysis to analyze the impact of government expenditure on poverty.

5.9.4 Cost-effectiveness data collection:

Health service costing data including capital costs, consumables, salaries etc. will be collected by careful review of health facility records and through consultation with administration staff. Costs to the community will be collected using an interviewer administered questionnaire recently developed by a GMP PhD student.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 3 months and 5 years at enrolment.
2. Informed consent obtained from parents or legal guardians.
3. No current participation in another malaria intervention trial.

Exclusion Criteria:

1. Previous adverse reaction to treatment with SP or amodiaquine. If this is unknown, then a history of allergic reaction to any drug.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14000 (Actual)
Dates: Start 2006-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Malaria incidence (the number of OPD attendances with clinical malaria that meet the case definitions as indicated below during the surveillance period ) and the number of hospital admissions with malaria during the surveillance period. | during malaria transmission period
Cost-effectiveness of the delivery system. | during the study period

SECONDARY OUTCOMES:
Coverage of IPTC | During the study period
the proportion of children who received three IPT courses on schedule; | during the study period
the proportion of children who received partial or off-schedule IPT courses | during the study period
the proportion of children with no IPT. | during the study period
Unit cost of delivery per fully adherent child. | during the study period
Incremental cost-effectiveness ratio for each systems of delivery. | During the study period
Mean Hb (g/dl) | at the end of malaria transmission
Prevalence of malaria parasitaemia | At the end of the malaria transmission season

CONTACTS AND LOCATIONS:
Overall Officials: Kalifa Bojang, MD, Principal Investigator — MRC Laboratories, The Gambia
Locations (1):
- MRC Laboratories, Banjul, The Gambia

REFERENCES:
- [Derived] Bojang KA, Akor F, Conteh L, Webb E, Bittaye O, Conway DJ, Jasseh M, Wiseman V, Milligan PJ, Greenwood B. Two strategies for the delivery of IPTc in an area of seasonal malaria transmission in the Gambia: a randomised controlled trial. PLoS Med. 2011 Feb 1;8(2):e1000409. doi: 10.1371/journal.pmed.1000409. PMID 21304921